CLINICAL TRIAL: NCT01728805
Title: Open-Label, Multi-Center, Randomized Study of Anti-CCR4 Monoclonal Antibody KW-0761 (Mogamulizumab) Versus Vorinostat in Subjects With Previously Treated Cutaneous T-Cell Lymphoma
Brief Title: Study of KW-0761 Versus Vorinostat in Relapsed/Refractory CTCL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0761-010
Record Dates: First submitted 2012-10-25; First posted 2012-11-20 (Estimated); Results first posted 2019-04-11 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Cutaneous T-Cell Lymphoma
Keywords: Cutaneous T-Cell Lymphoma (CTCL); myocis fungoides (MF); Sezary Syndrome (SS)
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Sezary Syndrome | interventions — mogamulizumab; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KW-0761 (Experimental): anti-CCR4 monoclonal antibody KW-0761 (mogamulizumab)
  Interventions: Biological: KW-0761
- Vorinostat (Active Comparator): vorinostat 400 mg once daily
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Biological: KW-0761 — 1.0 mg/kg weekly x 4 in cycle 1 then every other week until progression
  Other Names: mogamulizumab; POTELIGEO®
  Arms: KW-0761
Drug: Vorinostat
  Other Names: 400 mg orally daily; ZOLINZA®
  Arms: Vorinostat

SUMMARY:
The purpose of this study is to compare the progression free survival of KW-0761 versus vorinostat for subjects with relapsed or refractory CTCL.

DETAILED DESCRIPTION:
Phase 3 randomized study to compare the progression free survival of subjects with relapsed/refractory CTCL who receive KW-0761 versus those who receive vorinostat. Subjects who progress on vorinostat will be allowed to cross over to KW-0761 upon progression.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 years of age at the time of enrollment, except in Japan where subjects must be ≥ 20 years of age at the time of enrollment
* Histologically confirmed diagnosis of mycosis fungoides (MF) or Sezary Syndrome (SS)
* Stage IB, II-A, II-B, III and IV
* Subjects who had failed at least one prior course of systemic therapy. Psoralen plus ultraviolet light therapy (PUVA) is not considered to be a systemic therapy
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 1 at study entry
* Resolution of all clinically significant toxic effects of prior cancer therapy to grade ≤1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI-CTCAE, v.4.0)
* Adequate hematological, renal and hepatic function
* Subjects previously treated with anti-CD4 antibody or alemtuzumab were eligible provided their CD4+ cell counts were ≥ 200/mm3
* Subjects with mycosis fungoides (MF) and a known history of non-complicated staphylococcus infection/colonization were eligible provided they continued to receive stable doses of prophylactic antibiotics
* Women of childbearing potential (WOCBP) must have had a negative pregnancy test within 7 days of receiving study medication
* WOCBP and male subjects as well as their female partners of childbearing potential must have agreed to use effective contraception throughout the study and for 3 months after the last dose of KW-0761

Exclusion Criteria:

* Prior treatment with KW-0761 or vorinostat.
* Large cell transformation. However, subjects with a history of LCT but without current aggressive disease and no current evidence of LCT on pathology in skin and lymph nodes would be eligible.
* Diagnosed with a malignancy in the past two years. However, subjects with non-melanoma skin cancers, melanoma in situ, localized cancer of the prostate with current PSA of <0.1 ng/mL, treated thyroid cancer or cervical carcinoma in situ or ductal/lobular carcinoma in situ of the breast within the past two years could enroll as long as there was no current evidence of disease.
* Clinical evidence of central nervous system (CNS) metastasis.
* Psychiatric illness, disability or social situation that would have compromised the subject's safety or ability to provide consent, or limited compliance with study requirements.
* Significant uncontrolled intercurrent illness
* Known or tested positive for human immunodeficiency virus (HIV), human T-cell leukemia virus (HTLV-1), hepatitis B or hepatitis C.
* Active herpes simplex or herpes zoster. Subjects on prophylaxis for herpes who started taking medication at least 30 days prior to study entry, and had no active signs of active infection, and whose last active infection was more than 6 months ago, could enter the study, and should have continued to take the prescribed medication for the duration of the study.
* Experienced allergic reactions to monoclonal antibodies or other therapeutic proteins.
* Known active autoimmune disease were excluded. (For example, Grave's disease; systemic lupus erythematosus; rheumatoid arthritis; Crohn's disease; psoriasis).
* Was pregnant (confirmed by beta human chorionic gonadotrophin [β-HCG]) or lactating.
* History of allogeneic transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2021-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri O. Grebennik, MD, Study Director — Kyowa Kirin, Inc.
Locations (73):
- United States (34):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Banner MD Anderson, Gilbert, Arizona
  - City of Hope National Medical Center, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford Medical Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Yale University School of Medicine - Yale Cancer Center, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - The Winship Cancer Institute (Emory University), Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Tulane University Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Department of Medicine, Section of Hem/Onc, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Universal Dermatology, PLLC, Fairport, New York
  - Columbia Presbyterian, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester School of Medicine, Rochester, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - M.D.Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Parkville Cancer Clinical Trials Unit, Melbourne, Victoria
- Aarhus University Hospital, Aarhus, Denmark
- France (4):
  - CHU de Nantes, Nantes
  - Hôpital Saint Louis, Paris
  - CHU Bordeaux - Hopital Haut-Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (2):
  - University Medical Centre Mannheim, Mannheim
  - University Hospital Muenster, Münster
- Italy (2):
  - Institute of Hematology and Oncology Lorenzo e Ariosto Seràgnoli, University of Bologna, Bologna
  - Universita degli Studi di Torino, Turin
- Japan (19):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gunma University Hospital, Maebashi, Gunma
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Imamura Bun-in Hospital, Kagoshima, Kagoshima-ken
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nankoku-shi, Kochi
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Shinshu University Hospital, Matsumoto-shi, Nagano
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Tokyo Metropolitan Tama Medical Center, Fuchu-shi, Tokyo
  - Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- Leiden University Medical Center - Leids Universitair Medisch Centrum (LUMC), Leiden, Netherlands
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca
- University Hospital Zurich, Zurich, Switzerland
- United Kingdom (3):
  - The Christie Hospital Foundation NHS Trust, Manchester, Greater Manchester
  - University Hospital Birmingham, Birmingham
  - Guys & St. Thomas NHS Trust, London

REFERENCES:
- [Derived] Ortiz Romero PL, Kim YH, Molloy K, Quaglino P, Scarisbrick J, Thornton S, Sandilands K, Dent JE, Nixon A, Williams A, Shinohara MM. Health-related quality of life in cutaneous T-cell lymphoma: A post hoc analysis of a phase 3 trial in mycosis fungoides and Sezary syndrome. J Eur Acad Dermatol Venereol. 2025 Apr;39(4):833-845. doi: 10.1111/jdv.20357. Epub 2024 Sep 24. PMID 39315857
- [Derived] Kim YH, Bagot M, Pinter-Brown L, Rook AH, Porcu P, Horwitz SM, Whittaker S, Tokura Y, Vermeer M, Zinzani PL, Sokol L, Morris S, Kim EJ, Ortiz-Romero PL, Eradat H, Scarisbrick J, Tsianakas A, Elmets C, Dalle S, Fisher DC, Halwani A, Poligone B, Greer J, Fierro MT, Khot A, Moskowitz AJ, Musiek A, Shustov A, Pro B, Geskin LJ, Dwyer K, Moriya J, Leoni M, Humphrey JS, Hudgens S, Grebennik DO, Tobinai K, Duvic M; MAVORIC Investigators. Mogamulizumab versus vorinostat in previously treated cutaneous T-cell lymphoma (MAVORIC): an international, open-label, randomised, controlled phase 3 trial. Lancet Oncol. 2018 Sep;19(9):1192-1204. doi: 10.1016/S1470-2045(18)30379-6. Epub 2018 Aug 9. PMID 30100375

RESULTS

PARTICIPANT FLOW:
Groups:
- Vorinostat: vorinostat 400 mg once daily
  Vorinostat
- Vorinostat Original Then Crossover to KW-0761: Subjects who were randomized to vorinostat could be crossed over to receive mogamulizumab upon disease progression and with permission from the Medical Monitor.
Period: Randomization Period
Arm/Group | KW-0761 | Vorinostat | Vorinostat Original Then Crossover to KW-0761
Started | 186 | 186 | 0
Completed | 186 | 186 | 0
Not Completed | 0 | 0 | 0
Period: Crossover Period
Arm/Group | KW-0761 | Vorinostat | Vorinostat Original Then Crossover to KW-0761
Started | 0 | 0 | 136
Completed | 0 | 0 | 136
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KW-0761 | Vorinostat | Total
Number analyzed (Participants) | 186 | 186 | 372
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 99 | 89 | 188
  >=65 years | 87 | 97 | 184
Age, Continuous [Mean (Full Range); unit: years] | 62.8 [25 to 101] | 63.3 [25 to 89] | 63.0 [25 to 101]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 79 | 156
  Male | 109 | 107 | 216
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 125 | 135 | 260
  Race/Ethnicity: Other | 37 | 26 | 63
  Race/Ethnicity: Not Reported | 24 | 25 | 49
Region of Enrollment [Number; unit: participants]
  Netherlands | 0 | 2 | 2
  United States | 98 | 103 | 201
  Japan | 9 | 6 | 15
  Denmark | 1 | 2 | 3
  Italy | 14 | 12 | 26
  United Kingdom | 16 | 14 | 30
  France | 23 | 24 | 47
  Australia | 9 | 7 | 16
  Switzerland | 2 | 2 | 4
  Germany | 5 | 6 | 11
  Spain | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression was defined as follows, based on Olsen (2011):
  * Lymph nodes: ≥ 50% increase in SPD from baseline of lymph nodes, any new node > 1.5 cm in the long axis or > 1 cm in the short axis if 1-1.5 cm in the long axis that is proven to be N3 histologically, or > 50% increase from nadir in SPD of lymph nodes in those with PR
  * Skin: ≥ 25% increase in skin disease from baseline, new tumors (T3) in patients with T1, T2 or T4 only skin disease, or in those with CR or PR, increase of skin score of greater than the sum of nadir plus 50% baseline score
  * Blood: B0 to B2, > 50% increase from baseline and at least 5,000 neoplastic cells/μL36, or > 50% increase from nadir and at least 5,000 neoplastic cells/μL
  * Viscera: > 50% increase in size (SPD) of any organs involved at baseline, new organ involvement, or > 50% increase from nadir in the size (SPD) of any previous organ involvement in those with PR
Time Frame: From date of randomization at every visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | KW-0761 | Vorinostat
Number analyzed (Participants) | 186 | 186
percentage of subjects
  Rate (%) of Being Alive w/o Progression at 6 mos. | 55.3 [47.1 to 62.6] | 28.8 [21.6 to 36.3]
  Rate (%) of Being Alive w/o Progression at 12 mos. | 38.3 [30.2 to 46.4] | 15.3 [9.5 to 22.3]
  Rate (%) of Being Alive w/o Progression at 18 mos. | 28.0 [19.8 to 36.8] | 7.2 [2.7 to 14.5]
  Rate (%) of Being Alive w/o Progression at 24 mos. | 14.1 [6.4 to 24.8] | 7.2 [2.7 to 14.5]
  Rate (%) of Being Alive w/o Progression at 30 mos. | 4.7 [0.5 to 17.7] | 7.2 [2.7 to 14.5]

2. Secondary Outcome: Overall Response Rate
Description: The ORR was defined as the count of subjects who had a confirmed CR or PR, defined as documented CR or PR per Global Composite Response Score that was confirmed by a subsequent observation at least 4 weeks later. Overall Response Rate was determined based on the response in all compartments (lymph nodes, skin, peripheral blood, and viscera), referencing Olsen, 2011 as follows: Complete Response (CR) = complete disappearance of all clinical evidence of disease; Partial Response (PR) = regression of measurable disease; Stable Disease (SD) = failure to attain CR, PR, or PD; Progressive Disease (PD) = PD in any compartment; Relapse = recurrence of disease in prior CR in any compartment.
Time Frame: at the end of cycle 1 (26-28 days), and then every other cycle in Year 1 (cycle 3, 5, 7, 9, 11, 13), and every 16 weeks (cycle 17, 21, etc.) in Year 2 and beyond until progression up to 36 months
Population: The total number of patients analyzed are further broken out by disease type [mycosis fungoides (MF) and Sezary Syndrome (SS)]
Measure: Count of Participants; unit: Participants
Arm/Group | KW-0761 | Vorinostat
Number analyzed (Participants) | 186 | 186
Participants
  All Subjects ORR (confirmed CR + PR) | 52 | 9
  Disease Type = MF ORR (confirmed CR + PR): number analyzed (Participants) | 105 | 99
  Disease Type = MF ORR (confirmed CR + PR) | 22 | 7
  Disease Type = SS ORR (confirmed CR + PR): number analyzed (Participants) | 81 | 87
  Disease Type = SS ORR (confirmed CR + PR) | 30 | 2

3. Secondary Outcome: Quality of Life (QoL) Assessment - Skindex-29 Symptoms Scale Score
Description: * Skindex-29 rates 29 items assessing 3 domains (emotions, symptoms, & functioning) on a linear scale from 0 (never) to all the time (100). Higher scores = higher impact of skin disease.
  * FACT-G rates 27 items in 4 domains (physical well-being, social/family well-being, emotional well-being, functional well-being) on a 5-point scale from 0 (not at all) to 4 (very much). Higher scores = better QoL.
  * EuroQoL lvl 3 (Eq-5D-3L) rates mobility, self-care, usual activities, pain/discomfort and anxiety/depression on 3 levels - no problems, some problems, extreme problems. Score is calculated using a set of item weights to derive a single score ranging from -0.109 to 1, with 1 representing full health.
  LS mean (and 95% CI) of the overall change from baseline across time points through 6-month assessment (including End of Cycles 1, 3, and 5 time points only) are calculated from MMRM with treatment, disease type, disease stage, and region as fixed effects and baseline score as a covariate.
Time Frame: Cycle 1, 3, and 5
Population: The number of subjects analyzed in each row is the number of subjects with values at baseline and the specified post-baseline timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | KW-0761 | Vorinostat
Number analyzed (Participants) | 186 | 186
score on a scale
  Skindex-29 Across 6-month Assessment: number analyzed (Participants) | 162 | 171
  Skindex-29 Across 6-month Assessment | -12.6 [-15.94 to -9.29] | -6.0 [-9.39 to -2.52]
  FACT-G Across 6-month Assessment: number analyzed (Participants) | 167 | 177
  FACT-G Across 6-month Assessment | 4.6 [2.14 to 7.04] | -2.3 [-4.84 to 0.21]
  EQ-5D-3L Across 6-month Assessment: number analyzed (Participants) | 169 | 174
  EQ-5D-3L Across 6-month Assessment | 0.06 [0.028 to 0.085] | 0.02 [-0.008 to 0.052]

4. Secondary Outcome: Pruritis Evaluation
Description: The Itchy QoL is a validated pruritus specific quality of life instrument. It includes 22 pruritus-specific questions covering three major domains: symptoms, functioning, and emotions. The scale ranges from Never (1) to All The Time (5). The subscale scores consist of the average of the responses to the items in a given subscale. The overall score is the average of the responses to all items. Higher Itchy QoL scores indicate worse quality of life.
  LS mean (and 95% CI) of the overall change from baseline across time points through 6-month assessment (including End of Cycles 1, 3, and 5 time points only) are calculated from MMRM with treatment, disease type, disease stage, and region as fixed effects and baseline score as a covariate.
Time Frame: Cycle 1, 3, and 5
Population: The number of participants analyzed were subjects with values at baseline and post-baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | KW-0761 | Vorinostat
Number analyzed (Participants) | 166 | 175
score on a scale | -0.5 [-0.66 to -0.39] | -0.4 [-0.52 to -0.24]

ADVERSE EVENTS:
Time Frame: All subjects were assessed regularly for potential occurrence of adverse events from the time of signing the informed consent until 90 days after the last dose or initiation of alternative therapy, whichever came first, assessed up to 36 months.
Description: The following tables are based on the safety analysis set (all subjects who received at least one dose, even a partial dose, of the assigned study agent). Two subjects randomized to the mogamulizumab arm withdrew consent prior to receiving the first dose subsequently did not receive study treatment, bringing the number from 186 to 184.
  One subject crossed over from vorinostat to mogamulizumab but discontinued before receiving treatment, bringing the number from 136 to 135.
Arm/Group | KW-0761 | Vorinostat | Vorinostat Original Then Crossover to KW-0761
All-Cause Mortality (participants affected / at risk) | 40/184 | 47/186 | 32/135
Serious Adverse Events (participants affected / at risk) | 69/184 | 46/186 | 40/135
Other Adverse Events (participants affected / at risk) | 178/184 | 182/186 | 128/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KW-0761 (N=184) | Vorinostat (N=186) | Vorinostat Original Then Crossover to KW-0761 (N=135)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Anaemia Haemolytic Autoimmune (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Left Ventricular Hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Lens Dislocation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal Vein Occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Gastric Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large Intestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip Swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 1 (1)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device Failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 4 (4) | 1 (1) | 0 (0)
Facial Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
General Physical Health Deterioration (General disorders) | 1 (1) | 1 (2) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Localised Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 2 (3)
Pyrexia (General disorders) | 8 (9) | 1 (1) | 2 (5)
Autoimmune Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatocellular Injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Contrast Media Allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthritis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atypical Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 5 (5) | 6 (6) | 3 (3)
Cytomegalovirus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterovirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epstein-Barr Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes Simplex (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Otitis Externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Periorbital Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis Jiroveci Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2) | 2 (2)
Pneumonia Influenzal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Legionella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (4) | 5 (5) | 2 (2)
Sepsis Syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic Embolus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Staphylococcal Abscess (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Staphylococcal Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 2 (3) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 2 (3) | 0 (0) | 1 (1)
Blood Alkaline Phospatase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Infected Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Mycosis Fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 1 (1)
Depressed Level of Consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Miller Fisher Syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Motor Dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema Genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Drug Eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Social Stay Hospitalization (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Cardiac Pacemaker Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Air Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic Stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KW-0761 (N=184) | Vorinostat (N=186) | Vorinostat Original Then Crossover to KW-0761 (N=135)
Anaemia (Blood and lymphatic system disorders) | 20 (35) | 18 (20) | 9 (10)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 7 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 21 (34) | 56 (83) | 11 (48)
Dry Eye (Eye disorders) | 7 (7) | 11 (11) | 0 (0)
Vision Blurred (Eye disorders) | 8 (9) | 12 (14) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 7 (8) | 21 (24) | 7 (7)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 11 (12) | 0 (0)
Constipation (Gastrointestinal disorders) | 23 (27) | 34 (37) | 15 (15)
Diarrhoea (Gastrointestinal disorders) | 45 (62) | 114 (180) | 22 (33)
Dry Mouth (Gastrointestinal disorders) | 4 (4) | 17 (17) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 11 (11) | 0 (0)
Nausea (Gastrointestinal disorders) | 29 (38) | 78 (99) | 10 (13)
Stomatitis (Gastrointestinal disorders) | 10 (16) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (13) | 23 (33) | 0 (0)
Asthenia (General disorders) | 10 (12) | 25 (32) | 11 (18)
Chills (General disorders) | 13 (17) | 14 (15) | 8 (8)
Fatigue (General disorders) | 44 (55) | 69 (75) | 14 (19)
Oedema Peripheral (General disorders) | 27 (32) | 26 (37) | 13 (16)
Pyrexia (General disorders) | 26 (28) | 11 (11) | 17 (25)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 9 (12)
Folliculitis (Infections and infestations) | 14 (19) | 4 (4) | 13 (18)
Nasopharyngitis (Infections and infestations) | 13 (19) | 16 (23) | 9 (12)
Oral Candidasis (Infections and infestations) | 10 (10) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 17 (28) | 10 (15) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 20 (28) | 8 (9) | 12 (22)
Urinary Tract Infection (Infections and infestations) | 13 (17) | 14 (20) | 7 (8)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 8 (8)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 59 (83) | 0 (0) | 47 (55)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 12 (13)
Aspartate Aminotransferase Increased (Investigations) | 7 (8) | 12 (19) | 13 (15)
Blood Creatinine Increased (Investigations) | 6 (9) | 52 (58) | 0 (0)
Platelet Count Decreased (Investigations) | 4 (6) | 19 (22) | 0 (0)
Weight Decreased (Investigations) | 11 (15) | 32 (35) | 9 (9)
Weight Increased (Investigations) | 15 (17) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 14 (14) | 45 (49) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 15 (29) | 13 (28) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (15) | 11 (16) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (14) | 11 (17) | 15 (17)
Back Pain (Musculoskeletal and connective tissue disorders) | 17 (20) | 9 (10) | 10 (13)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 10 (11) | 29 (49) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (14) | 8 (8) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 13 (17) | 10 (16) | 13 (13)
Dizziness (Nervous system disorders) | 12 (13) | 19 (20) | 8 (11)
Dysgeusia (Nervous system disorders) | 8 (8) | 55 (59) | 0 (0)
Headache (Nervous system disorders) | 23 (35) | 27 (32) | 17 (32)
Paraesthesia (Nervous system disorders) | 5 (5) | 14 (16) | 8 (10)
Depression (Psychiatric disorders) | 10 (10) | 6 (6) | 0 (0)
Insomnia (Psychiatric disorders) | 16 (16) | 14 (14) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 16 (19) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (14) | 7 (8) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 5 (7) | 7 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (13) | 35 (35) | 9 (9)
Drug Eruption (Skin and subcutaneous tissue disorders) | 44 (77) | 1 (2) | 35 (54)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 7 (12)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 11 (15)
Hypertension (Vascular disorders) | 17 (38) | 25 (28) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/05/NCT01728805/Prot_002.pdf
  • Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT01728805/SAP_001.pdf